CLINICAL TRIAL: NCT00860496
Title: A Phase I, Open Label, Fixed-Sequence Study to Estimate the Effect of Tacrolimus and Cyclosporine on the Pharmacokinetics of CP-690,550 in Healthy Volunteers
Brief Title: A Phase I Open-Label Study of the Effects of Tacrolimus and Cyclosporine on CP-690,555 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A3921020
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2009-08-13 (Estimated); Status verified 2009-08

CONDITIONS: Healthy Volunteers
Keywords: Immunosuppression, JAK3 inhibitor, calcineurin inhibitors, tacrolimus, cyclosporine, pharmacokinetics, safety, tolerability
MeSH Terms: interventions — tofacitinib; Tacrolimus; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Treatment Arm 1 will receive one single dose of CP-690,550 on Day 1, Tacrolimus on Days 1-8, and one single dose of CP-690,550 on Day 8.
  Interventions: Drug: CP- 690,550 and Tacrolimus
- 2 (Other): Treatment Arm 2 will receive one single dose of CP-690,550 on Day 1, Cyclosporine on Days 1-6, and one single dose of CP-690,550 on Day 6.
  Interventions: Drug: CP- 690,550 and Cyclosporine

INTERVENTIONS:
Drug: CP- 690,550 and Tacrolimus — 10 mg, single dose of CP-690,550 on Day 1 5 mg, every 12 hours of Tacrolimus on Days 1-8 10 mg, single dose of CP-690,550 on Day 8
  Arms: 1
Drug: CP- 690,550 and Cyclosporine — 10 mg, single dose of CP-690,550 on Day 1 200 mg, every 12 hours of Cyclosporine on Days 1-6 10 mg, single dose of CP-690,550 on Day 6
  Arms: 2

SUMMARY:
A new immunosuppressive drug, based on the inhibition of important enzymes in the immune system, called JAK, is being developed by Pfizer to prevent transplant rejection. Since many treatments for transplant rejection may be administered together, this research study will analyze the effects of common transplant rejection therapies, Tacrolimus and Cyclosporine, on the JAK inhibitor, CP-690,550.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males between 21 and 55 years, inclusive.
* Healthy females of non-childbearing potential between 21 and 55 years, inclusive.
* Total body weight greater than 132 pounds.

Exclusion Criteria:

* Evidence or history of clinically significant disease
* Females of childbearing potential

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Effect of multiple dose Tacrolimus and Cyclosporine on the pharmacokinetics of a single oral dose of CP-590,550 in healthy volunteers | 9 days

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of a single oral dose of CP-690,550 when co-administered with Tacrolimus or Cyclosporine | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921020&StudyName=A%20Phase%20I%20Open-Label%20Study%20of%20the%20Effects%20of%20Tacrolimus%20and%20Cyclosporine%20on%20CP-690%2C555%20in%20Healthy%20Volunteers